CLINICAL TRIAL: NCT05426187
Title: Long Term Follow-up of Immunological Pattern and Pregnancy Outcomes in Women Previously Enrolled in a Phase 1b Clinical Trial With the PRIMVAC Placental Malaria Candidate Vaccine
Brief Title: Follow-up of Immunological Pattern and Pregnancy Outcomes in Women Previously Received Placental Malaria Vaccine
Acronym: PRIMVACLongT
Status: Active, not recruiting | Type: Observational
Sponsor: Groupe de Recherche Action en Sante (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); European Vaccine Initiative (Other)
Responsible Party: Sponsor
Other Study IDs: PRIMVAC Long Term study
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Malaria in Pregnancy
Keywords: vaccine; nulligravid; immunology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood smear dried blood spot venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Women who received the PRIMVAC Vaccine or Placebo during the phase 1b trial in Burkina Faso
- Group 2: Women of the same age and nulligravid who did not participate in the phase 1b trial
- Group 3: Women of the same age and primigravid who did not participate in the phase 1b trial

SUMMARY:
Study Population: Participants of the previous PRIMVAC vaccine trial and women aged 18 to 35 years

Sample Size: 90

Study duration: 21 months

Subject duration: 12 months if pregnancy doesn't occurred. In case of pregnancy, the participant will be followed up until the delivery.

Study Design: Long term observational study comparing the immunology trend of 3 groups of i) women who received the PRIMVAC Vaccine or Placebo during the phase 1b trial in Burkina Faso; ii) women of the same age and nulligravid who did not participate in the phase 1b trial iii) women of the same age and primigravid who did not participate in the phase 1b trial

Co Primary objectives

* To assess the dynamics of humoral immune response to the vaccine antigen during long term follow up of the study participants
* To evaluate the functional durability of the humoral immune responses of women who participated in the phase 1b vaccine trial compared to women of the same age

Secondary objectives

* To assess the cellular immune response during the follow-up period
* To assess the incidence of clinical malaria on study participants
* To assess the prevalence of Placental Malaria in study participants and adverse outcomes such as maternal anemia, low birth weight, stillbirth and prematurity.

DETAILED DESCRIPTION:
It is a long-term observational study comparing the immunology trend of 3 groups of women:

* Women who received the PRIMVAC Vaccine or Placebo during the phase 1b trial in Burkina Faso
* Women of the same age and nulligravid who did not participate in the phase 1b trial
* Women of the same age and primigravid who did not participate in the phase 1b trial

The proposed cohort study will build on the previous phase 1b study which was conducted within the health district of Saponé (ClinicalTrials.gov Identifier: NCT02658253). The enrolment and follow up of the subjects will last 12 months. Pregnancy which occurred during the follow up period will monitored until the delivery. An additional six months is necessary for sample analysis in the laboratory, the data analysis and the preparation of reports and publications.

ELIGIBILITY:
Inclusion Criteria:

* Any participant of the previous PRIMVAC vaccine phase Ib trial
* Nulligravid and primigravid women aged 18-35 years
* Residing in study region and environs
* Available and willing to participate in follow-up for the duration of study
* Participant who accept blood sample collection
* Appear to be in generally good health based on clinical and laboratory investigation
* Signed informed consent

Exclusion Criteria:

* Participants who refused to sign informed consent
* Use of an investigational or non-registered drug or vaccine other than the previous study vaccine
* Chronic administration of immunosuppressants or other immune-modifying drugs
* Confirmed or suspected immunosuppressive or immunodeficient condition
* Confirmed or suspected autoimmune disease
* Simultaneous participation in any interventional clinical trial
* Women of control groups with positif pregnancy test at the enrolment

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Placental malaria concern only the women
Study Population: Women who received the PRIMVAC Vaccine or Placebo during the phase 1b trial in Burkina Faso. Women of the same age and nulligravid who did not participate in the phase 1b trial. Women of the same age and primigravid who did not participate in the phase 1b trial.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer of antibodies | month 0
  Level of total Immunoglobin (IgG) and the level of the isotypic subtypes (IgG1, IgG2, IgG3, IgG4)
Geometric mean titer of antibodies | month 6
  Level of total Immunoglobin (IgG) and the level of the isotypic subtypes (IgG1, IgG2, IgG3, IgG4)
Geometric mean titer of antibodies | month 12
  Level of total Immunoglobin (IgG) and the level of the isotypic subtypes (IgG1, IgG2, IgG3, IgG4)
Cross-reactivity against different VAR2CSA variants expressed on the surface of erythrocytes parasitized by various strains of Plasmodium falciparum by flow cytometry | month 0
  VAR2CSA variants
Percentage of binding inhibitory activity using various VAR2CSA expressing strains by CSA-binding inhibition assay (BIA) at different timepoints during the twelve months of follow up. | month 0
  binding inhibitory activity

CONTACTS AND LOCATIONS:
Overall Officials: Alphonse Ouedraogo, MD, PhD, Principal Investigator — Groupe de Recherche Action en Sante
Locations (1):
- Groupe de Recherche Action en Santé, Ouagadougou, Burkina Faso

IPD SHARING:
Plan to Share IPD: No